CLINICAL TRIAL: NCT02118025
Title: Prospective Randomized Comparison of Coronary Bypass Grafting With Minimal Extracorporeal Circulation System (MECC) Versus Off-pump Coronary Surgery. New Insights Into Inflammatory Cytokines.
Brief Title: Coronary Bypass Grafting With Minimal Extracorporeal Circulation System Versus Off-pump Coronary Surgery
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: MECC-1; MECC-1 (Other: MECC-1)
Record Dates: First submitted 2014-03-25; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: Off-pump bypass graft surgery; Mini extracorporeal circulation bypass surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass, Off-Pump

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Off-pump coronary artery bypass graft: Patients operated on with off-pump coronary artery bypass graft, beating heart surgery.
  Interventions: Procedure: Off-pump coronary artery bypass graft
- Mini extracorporeal circulation bypass: Patients operated on with mini extracorporeal circulation bypass. A modified extracorporeal system.
  Interventions: Procedure: Mini extracorporeal circulation bypass

INTERVENTIONS:
Procedure: Off-pump coronary artery bypass graft — Patients operated with the heart beating, without heart arrest.
  Groups: Off-pump coronary artery bypass graft
Procedure: Mini extracorporeal circulation bypass — Patients operated with a modified extracorporeal circulation system
  Groups: Mini extracorporeal circulation bypass

SUMMARY:
The investigators aimed to evaluate the clinical results and the inflammatory response of the minimal extracorporeal circulation system (MECC) Compared with off-pump coronary revascularization (OPCABG).

This is a randomized and prospective study in 230 patients with indications for coronary surgery, with 113 patients in the OPCABG group and 117 in the MECC group. The endpoints were the clinical and biochemical results, intra-operative outcomes and the determination of 19 inflammatory circulating markers, 17 of them for the first time analyzed comparing both techniques.

ELIGIBILITY:
Inclusion Criteria:

* Indication for coronary surgery established on the basis of current published guidelines

Exclusion Criteria:

* Documented preoperative systemic proinflammatory status and/or steroid administration within 6 months before surgery.
* Coexistence of a cardiomyopathy different than coronary artery disease that precise surgical treatment.
* Left ventricle ejection fraction of 40% or less.
* Treatment with erythropoietin (EPO) three months before the intervention
* Hematocrit less than 35% the day prior to the procedure
* Redo surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 230 patients with indication for coronary surgery established on the basis of current published guidelines. All patients provided written consent to enter the study.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2006-01; Primary Completion 2008-11 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes | within the first 30 days (plus or minus 3 days) after surgery
  Number of Participants with Adverse Events, e.g, renal failure, atrial fibrillation, acute myocardial infarct, stroke, redo surgery, death.

SECONDARY OUTCOMES:
Determination of increase over the first 48 hours of plasma levels of 19 circulating markers of inflammatory response. | Area Under the Concentration-Time Curve (AUC 0-48 hours)
  Determination of increase over the first 48 hours after the operation of plasma levels of 19 circulating markers of inflammatory response. The levels of inflammatory markers are measured in pg / mL and subsequently, the increase over the 48 hours is determined with the area under the curve.
Biochemical outcomes | Within the first 30 days (plus or minus 3 days) after surgery
  Changes in creatine kinase levels, troponin levels, glucose, leukocytes, platelets, hemoglobin and hematocrit levels. From basal point to 48 hours time after surgery.
Operative results | Within the first 30 days (plus or minus 3 days) after surgery
  Number of distal anastomosis.
Operative results | Within the first 30 days (plus or minus 3 days) after surgery
  Type of grafts used.
Operative results | Within the first 30 days (plus or minus 3 days) after surgery
  time until removal of mechanical respiratory support
Operative results | Within the first 30 days (plus or minus 3 days) after surgery
  Time at intensive care unit (days)
Operative results | Within the first 30 days (plus or minus 3 days) after surgery
  Total hospitalization time (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Permanyer E, Munoz-Guijosa C, Padro JM, Ginel A, Montiel J, Sanchez-Quesada JL, Vila L, Camacho M. Mini-extracorporeal circulation surgery produces less inflammation than off-pump coronary surgery. Eur J Cardiothorac Surg. 2020 Mar 1;57(3):496-503. doi: 10.1093/ejcts/ezz291. PMID 31651944